CLINICAL TRIAL: NCT02180386
Title: Effect of PlayStation Distraction on Children's Behavior and Pain in the Dental Setting
Brief Title: Effect of PlayStation Distraction in the Dental Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, Effect of PlayStation Distraction on Children's Behavior and Pain in the Dental Setting, Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UIC-ODP-3
Record Dates: First submitted 2014-06-27; First posted 2014-07-02 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Global Behaviour Measure
Keywords: Audiovisual distraction; Pediatric dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental group (Experimental): Patients will play a video game with Rimax® multimedia eyeglasses that occlude the environment partially during the second treatment visit.
  Interventions: Behavioral: Patients will play a video game with Rimax® multimedia eyeglasses that occlude the environment partially during the second treatment visit.

INTERVENTIONS:
Behavioral: Patients will play a video game with Rimax® multimedia eyeglasses that occlude the environment partially during the second treatment visit. — videogame can be considered as a method of distraction.

SUMMARY:
The aim of the study was to assess whether the behavior, anxiety, and dental pain of pediatric patients during dental treatment improves when a video game is played as method of distraction.

DETAILED DESCRIPTION:
global behavior Parental perception of patients' anxiety Patient's anxiety dental pain Heart Rate

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6-8 years.
* Patients who required a minimum of 2 visits for restorative treatment.

Exclusion Criteria:

* Patients with reduced audiovisual capabilities.
* Patients with psychological disorders.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Global behavior during the treatment | 14 days
  we will use the Frankl Scale

SECONDARY OUTCOMES:
Parental perception of patient's anxiety | 14 days
  we will use the Modified Corah Anxiety Scale Questionnaire
Self-reported anxiety during the treatment | 14 days
  we will use the Venham Picture Test
Dental pain during the treatment | 14 days
  We will use the Wong-Baker Faces Scale
Heart rate during the treatment measures in different time points | 14 days
  We will use the the pulse oximeter
Degree of acceptance of the distraction method by the pediatric patient | 14 days
  "Did you enjoy seeing the cartoon film during the dental visit?" (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Background] Ram D, Shapira J, Holan G, Magora F, Cohen S, Davidovich E. Audiovisual video eyeglass distraction during dental treatment in children. Quintessence Int. 2010 Sep;41(8):673-679. PMID 20657857
- [Background] El-Sharkawi HF, El-Housseiny AA, Aly AM. Effectiveness of new distraction technique on pain associated with injection of local anesthesia for children. Pediatr Dent. 2012 Mar-Apr;34(2):e35-8. PMID 22583875